CLINICAL TRIAL: NCT04813081
Title: The Evaluation of Free Gingival Graft Operations Around Implant or Teeth on Quality of Life: Parallel-controlled Prospective Clinical Trial
Brief Title: The Evaluation of Free Gingival Graft Operations Around Implant or Teeth on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Collaborators: Kutahya Health Sciences University (Other); Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Serap Karakış Akcan, Assistant professor doctor, University of Beykent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.AYD.0.00.00-480.2/184
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Patient Reported Outcome
Keywords: quality of life; graft

STUDY DESIGN:
Intervention Model Description: The participants were defined as two study groups: Test Group (TG) consists of patients have free gingival graft around dental implant patients and Control Group (CG) consists of patients have free gingival graft around the teeth.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free gingival graft around dental implant patients (Active Comparator): Test Group (TG) consists of patients have free gingival graft around dental implant patients
  Interventions: Procedure: Free Gingival Graft
- Free gingival graft around the teeth (Active Comparator): Control Group (CG) consists of patients have free gingival graft around the teeth.
  Interventions: Procedure: Free Gingival Graft

INTERVENTIONS:
Procedure: Free Gingival Graft — In the recipient area, a half-thickness flap with two vertical incision widths was removed with a horizontal incision with 15C blades from the mucogingival junction. The recipient site was determined such that one or two teeth or one tooth extends into the mesial and distal regions of the tooth. Muscle attachments were dissected and FGG was placed on recipient bed and non-resorbable monofilament sutures were used for fixing the four corners of the graft.

SUMMARY:
The purpose of this study is to evaluate the quality of life of patients who underwent FGG surgery around the natural tooth and as a second surgery after the implant operation, in comparison with general oral health assesment index(GOHAI).

DETAILED DESCRIPTION:
Thirty-two participants were included who were referred to the periodontology clinic suffering insufficient keratinized gingiva / mucosa deficiency around the implant and / or tooth/teeth. GOHAI-total and GOHAI psychological impact, functional limitation, pain and discomfort, behavioral impact subcategories were recorded at before and postoperative first week and 30th day. Also, satisfaction questionnaires, number of painkillers and visual analog scale values were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Teeth and implants with keratinized gingiva width <1 mm
* A healthy periodontal and peri-implant condition
* Patients who didn't have ever experience periodontal surgery had first oral surgery experience with dental FGG operation for the first time
* Patients who underwent implant surgery for the first oral surgery experience
* Maximum two teeth/implants on recipient area

Exclusion Criteria:

* Patients receiving any medication to disrupt wound healing
* Lactation or pregnancy
* Caries or defects on the tooth root surface
* Periapical lesion in the recipient area active periodontal disease
* Patients who have previously had periodontal or oral surgery experiences

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
General Oral Health Assesment Index (GOHAI) scores- intragroup comparisons change between from baseline to other follow-up times and intergroup comparisons all follow-up times | Baseline, postoperative 1., 2., 3., 4., 5., 6. and 7. days and first month.
  The questions that contains 12 items and that give subcategorized about functional limitations, pain and discomfort, psychological impacts, and behavioral impact.

SECONDARY OUTCOMES:
Age | baseline
  18-65 years

OTHER OUTCOMES:
Gender | baseline
  male, female
Keratinized gingival width (KGW) | baseline, first month
  the distance between the gingival margin and mucogingival junction from tooth/implant in operation area
Graft volume (GV) | during surgery
  graft vertical height X graft mesiodistal length X graft thickness
Surgery localization | baseline
  maxilla, mandible, anterior, posterior
Operation time | during surgery
  operation time between of first incision and last suture
Satisfaction questionnaires | first month
  A questionnaire designed by authors with 12 questions was used to assess patient satisfaction. Answers were either categorized as "positive" or "negative".
Visual Analog Scale (VAS) | postoperative 1., 2., 3., 4., 5., 6. and 7. days
  a 100-mm horizontal scale and classify the level of postoperative pain experience from 0 (no pain) to 100 (the worst pain ever experienced)
Painkiller consumption | postoperative 1., 2., 3., 4., 5., 6. and 7. days
  the total number of painkillers for each follow-up day

CONTACTS AND LOCATIONS:
Overall Officials: serap karakış akcan, phd, Study Director — Beykent University; berceste güler, phd, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Beykent University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Zucchelli G, Tavelli L, McGuire MK, Rasperini G, Feinberg SE, Wang HL, Giannobile WV. Autogenous soft tissue grafting for periodontal and peri-implant plastic surgical reconstruction. J Periodontol. 2020 Jan;91(1):9-16. doi: 10.1002/JPER.19-0350. Epub 2019 Oct 6. PMID 31461778
- [Result] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Result] McGuire MK, Scheyer ET, Gwaltney C. Commentary: incorporating patient-reported outcomes in periodontal clinical trials. J Periodontol. 2014 Oct;85(10):1313-9. doi: 10.1902/jop.2014.130693. Epub 2014 Jul 18. PMID 25034790
- [Result] Locker D, Matear D, Stephens M, Lawrence H, Payne B. Comparison of the GOHAI and OHIP-14 as measures of the oral health-related quality of life of the elderly. Community Dent Oral Epidemiol. 2001 Oct;29(5):373-81. doi: 10.1034/j.1600-0528.2001.290507.x. PMID 11553110
- [Result] Mei CC, Lee FY, Yeh HC. Assessment of pain perception following periodontal and implant surgeries. J Clin Periodontol. 2016 Dec;43(12):1151-1159. doi: 10.1111/jcpe.12618. Epub 2016 Nov 2. PMID 27554366